CLINICAL TRIAL: NCT06146777
Title: A Multicenter, Open, Prospective Study of Prognostic Value and Benefit From Adjuvant Immunotherapy of Stage III Papillary Renal Cell Carcinoma Based on Multi-classifier System
Brief Title: Multi-classifier System for Stratifying Stage III Papillary Renal Cell Carcinoma of Receiving Adjuvant Therapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jun-Hang Luo, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstSunYatSen20231101
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Papillary Renal Cell Carcinoma
Keywords: Papillary renal cell carcinoma; pembrolizumab; Adjuvant therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg on Day 1 of each 3-week cycle for up to 17 cycles.
  Interventions: Drug: Pembrolizumab
- Placebo (Placebo Comparator): Participants receive intravenous placebo on Day 1 of each 3-week cycle for up to 17 cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Intravenous infusion
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
  Arms: Pembrolizumab
Drug: Placebo — Intravenous infusion
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
The goal of this trial is to test whether patients with stage III papillary renal cell carcinoma (pRCC) could benefit from adjuvant therapy or not. The investigators invented a multi-classifier system that was successfully categorise patients with stage III pRCC into high-risk and low-risk groups. Here the investigators randomly assign classifier-defined high risk patients of stage III pRCC into adjuvant pembrolizumab group placebo group. Disease-free survival and overall survival are the end points of observation.

DETAILED DESCRIPTION:
kidney cancer represented 4.2% of all new cancer cases, and its incidence has been increasing. Over 90% of kidney cancer cases are renal cell carcinoma (RCC), which includes various subtypes with distinct histologic features, clinical courses, and responses to therapy. Clear cell renal cell carcinoma (ccRCC) and papillary renal cell carcinoma (pRCC) are the most common histologic subtypes of RCC, accounting for approximately 75% and 20% of all cases, respectively. Adjuvant pembrolizumab showed promising efficacy in ccRCC, however, whether high-risk pRCC patients could benefit from adjuvant pembrolizumab remain unknown.

Participants will be assigned to continue with the study treatment until any of the following occurs: the recurrence of the disease; the emergence of unacceptable adverse events (AEs); the presence of an intercurrent illness that precludes further administration of the treatment; the decision of the Investigator to withdraw the participant; noncompliance with the study treatment or procedural mandates; administrative reasons necessitating the discontinuation of treatment; or the completion of 17 treatment cycles (approximately one year), with each cycle 3 weeks long.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of pRCC
* With confirmed diagnosis of stage III pRCC
* Classified as high-risk by multi-classifier system
* With moderate/good Eastern Cooperative Oncology Group (ECOG) health rating (PS): 0-1 score.
* Receive radical operation for renal cancer with negative margin.
* Receive no anti-cancer treatment before primary surgery.
* The informed consent has been obtained from the patient.

Exclusion Criteria:

* Patients with Transcription factor enhancer 3(TFE3) or transcription factor EB (TFEB) translocation proven by cytogenetic analysis or by fluorescence in situ hybridization (FISH)
* Previously received neoadjuvant therapy
* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.
* Pregnant woman or lactating woman.
* With contraindication to receive pembrolizumab, such as had a prior solid organ transplant, has a known history of human immunodeficiency virus infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From the date of registration to up to 7 years
  Disease free survival (DFS) was defined as the time interval (in years) from the date of randomization to the first date of recurrence or occurrence of a secondary malignancy or death.

SECONDARY OUTCOMES:
Overall survival | From the date of registration to up to 7 years
  Overall survival (OS) was defined as the time from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hang Luo, M.D., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University